CLINICAL TRIAL: NCT06327191
Title: EMERGE Mothers and Kids: a Longitudinal Cohort Study of Mothers and Kids Enrolled in the Randomized Placebo Controlled Trial of Metformin in Women With GDM (EMERGE)
Brief Title: EMERGE Mothers and Kids
Status: Recruiting | Type: Observational
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Fidelma Dunne, Professor, National University of Ireland, Galway, Ireland
Other Study IDs: 23-CRFG-21; 23-CRFG-21 (Other: Clinical Research Facility Galway (CRFG) study number)
Record Dates: First submitted 2023-11-21; First posted 2024-03-25 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention as the study is observational. — No intervention as the study is observational.

SUMMARY:
The EMERGE Mothers and Kids study is a follow-up to the EMERGE trial of women with GDM (N=535) that aimed to determine the effect of the addition of metformin compared to placebo on insulin initiation rates, maternal weight gain and perinatal morbidity and mortality.

The primary objectives of the EMERGE Mothers and Kids follow up study are:

1. to determine whether treatment with metformin leads to a reduction in maternal disorders of glucose, metabolic syndrome, obesity, hypertension and lipids at up to 10 years post the index pregnancy;
2. to examine the impact of metformin on maternal anxiety, depression, quality of life and breast feeding duration;
3. to examine whether exposure to metformin leads to a reduction in obesity in the offspring at follow up;
4. to determine whether treatment with metformin during pregnancy, in women with GDM, leads to a reduction in adiposity in the offspring at follow up as measured by anthropometric measurements and sum of skinfolds.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the original EMERGE trial and consenting to further follow up.

Exclusion Criteria:

* EMERGE trial participants who did not provide consent for further follow up studies.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants only
Study Population: The population for this longitudinal cohort study is women who participated in the EMERGE randomised controlled trial and who consented to be contacted about further follow-up studies.
Sampling Method: Probability Sample
Enrollment: 321 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To assess if treatment of GDM with metformin during pregnancy compared to placebo reduces the risk of disorders of glucose metabolism at follow up.. | Up to 10 years post the index pregnancy
  This will be evaluated using a 75g oral glucose tolerance test (OGTT) and a haemoglobin A1c (HbA1c). Cutoffs for diabetes, imparied fasting gluocse and impaired glucose tolerance will be in line with the American Diabetes Association diagnostic criteria (ADA 2023).
To assess if treatment of GDM with metformin during pregnancy compared to placebo reduces the risk of metabolic syndrome. | Up to 10 years post the index pregnancy
  Metabolic syndrome is defined as the presence of >3 of the following risk factors (International Diabetetes Foundation 2009)
  * Fasting glucose >5.6 mmol/L or diagnosed diabetes
  * High density lipoprotein (HDL) cholesterol of <1.3 mmol/L or drug treatment for low HDL cholesterol
  * Triglyceride level of >1.7 mmol/L or drug treatment for elevated triglycerides
  * Waist circumference of >80cm
  * Hypertension with a blood pressure of > 130/85 mmHg or drug treatment for hypertension
To assess if treatment of GDM with metformin during pregnancy compared to placebo reduces rates of OW and OB at follow up. | Up to 10 years post the index pregnancy
  Definitions of overweight and obesity are a body mass index of >25 kg/m2 and >30 kg/m2, respectively.
To assess if treatment of GDM with metformin during pregnancy compared to placebo reduces the risk of hypertension. | Up to 10 years post the index pregnancy
  Hypertension is defined as a blood pressure of > 130 mmHg systolic or >80 mmHg diatolic (Whelton 2017).
To examine the associations of GDM diagnosis, sum of fasting, 1-hour, and 2-hour glucose z-scores after 75-g load, insulin sensitivity, and lipid levels at 24-32 weeks' gestation with lipid levels at up to 10 years postpartum. | Up to 10 years post the index pregnancy
  Lipid levels will be assessed by measuring a fasting sample and will be analysed using local assays.
To determine whether treatment with metformin during pregnancy, in women with GDM, leads to a reduction in adiposity in the offspring at follow up as measured by anthropometric measurements and sum of skinfolds. | Up to 10 years post the index pregnancy
  Obesity will be defined as a BMI of >95th percentile or BMI > 30 kg/m2 (whichever is lower) for children 2 years and older. Overweight will be defined as a BMI of >85th percentile.
  Weight for height gender specific growth charts will be used for children <2 years of age and a weight-for-height which is >95th centile will be considered obese. Overweight wil be defined as a BMI of >85th percentile.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No